CLINICAL TRIAL: NCT06652204
Title: Validation of the French Version of the Informal Caregiver Burden Assessment Questionnaire (QASCI) in Caregivers of Patients With COPD (VALQASCI)
Brief Title: Validation of the French Version of the QASCI in Caregivers of Patients With COPD
Acronym: VALQASCI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Collaborators: Centre Hospitalier des Pays de Morlaix (Other)
Responsible Party: Principal Investigator, BEAUMONT Marc, principal investigator, University Hospital, Brest
Other Study IDs: 29BRC24.0115 - VALQASCI
Record Dates: First submitted 2024-10-15; First posted 2024-10-22 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Caregiver
Keywords: validation of questionnaire; caregivers burnout; copd
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- caregivers of patients with COPD
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Caregivers must reply to the French version of the QASCI questionnaire, the ZBI (Zarit Burden Interview) questionnaire, HADS (Hospital Anxiety and Depression Scale), and WHOQOL-Bref (World Health Organization Quality of Life Instrument - Short Form). After 15 days, they wil reply to the French version of the QASCI questionnaire (to asse the reliability).

SUMMARY:
This study aims to validate the French version of the QASCI questionnaire, initially written and validated in Portuguese language by Hipolito et al., to assess caregiving burden in chronic obstructive pulmonary disease (COPD).

The realization of this validation is significant on several levels. First, since COPD is a systemic condition, it affects not only the lungs but also many other organs and systems in the body. It leads to various complications that go beyond respiratory symptoms, creating major challenges not only physically but also in terms of participation and involvement for patients and their caregivers. The lack of validated tools in French to specifically assess the quality of life of caregivers in this context represents a gap that this study seeks to fill.

This study is also justified by the fact that, although the QASCI has been validated in other languages and contexts, it is essential to linguistically and culturally adapt this tool for the French-speaking population. Validation in French is crucial to ensure the fidelity of the results obtained and the validity of the conclusions drawn from this instrument for caregivers of patients with COPD in France.

In summary, this study addresses a specific need by contributing to the prevention of pathologies among caregivers. It enhances early detection and support for caregivers of patients with COPD while paving the way for future research on this often-overlooked population.

DETAILED DESCRIPTION:
Beyond its respiratory component, COPD, being a systemic condition, leads to significant problems in various domains for patients. Dyspnea remains their main complaint, but these patients also experience impairments in physical capacity, nutritional status, and symptoms of anxiety and depression, which can limit their daily physical activity and reduce their quality of life, even their life expectancy.

As the disease progresses, patients become increasingly dependent on care, experiencing difficulties in performing activities of daily living (ADLs), and social isolation is often observed.

In this context, caregivers (usually a spouse or child) play a crucial role in supporting patients with ADLs, providing assistance with medical care and symptom management. Their presence is essential for facilitating and improving patients' adherence to COPD management behaviors, such as treatment compliance or increasing daily physical activity. Thus, their role in the healthcare system is fundamental, both as a link to medical teams and as support for the patient.

However, assuming the caregiver role can heavily impact the caregiver's physical, psychological, and social well-being. A survey in Spain reveals that many caregivers face health issues and experience reduced social, leisure, and professional activities due to their role. Additionally, they may feel helpless, anxious, depressed, and vulnerable to fatigue, incapacity, and/or burnout while trying to cope with the demands related to COPD. Other studies highlight the professional impact of caregiver status, with absences linked to this situation or decreased work effectiveness. This situation can be even more challenging for caregivers of patients with advanced COPD, who face higher risks of exacerbations, hospitalizations, and mortality compared to less severely affected patients.

It is therefore essential that healthcare professionals and paramedical staff who work with COPD patients and their caregivers have a tool to assess the burden on informal caregivers. To date, the only existing tool seems to be the QASCI questionnaire, drafted and validated in Portuguese by Hipólito et al. However, due to the language barrier, this tool cannot be used with French-speaking populations.

It is in this context that the present study finds its place, with the aim of establishing the validity and reliability of the French translation of the QASCI questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Being a caregiver of a relative with COPD (according to the GOLD criteria).
* Being 18 years old or older.
* The patient under the caregiver's care must be in stable condition (no exacerbations in the previous month).
* Being a family member of the patient or living with the patient.
* Being able to complete the French questionnaires.
* Non-opposition statement provided.

NON-INCLUSION CRITERIA

* Person under judicial protection (guardianship, curatorship, etc.)
* Refusal to participate
* The patient under the caregiver's care has experienced an exacerbation in the previous month
* The caregiver reports that the patient has cognitive impairments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Informal caregivers of patients with COPD
Sampling Method: Probability Sample
Enrollment: 224 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Validation of the translation of the long version of the QASCI questionnaire (measuring caregiver burden) from Portuguese to French after the translation-back translation stage. | baseline
  Responses to the QASCI questionnaire (32 items rated from 1 to 5 leading to an overall score and 7 subscores) and comparison with responses to the ZBI (Zarit Burden Interview), HADS (Hospital Anxiety and Depression Scale), and WHOQOL-Bref (World Health Organization Quality of Life Instrument - Short Form).

SECONDARY OUTCOMES:
Assess the reliability of the translation of the long version of the QASCI questionnaire. | baseline and at day 15
  Responses to the QASCI questionnaire (32 items rated from 1 to 5 leading to an overall score and 7 subscores) at Day 0 and Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Marc Beaumont, PhD, Principal Investigator — Centre Hospitalier des Pays de Morlaix
Locations (2):
- France (2):
  - Chu Brest, Brest
  - Centre hospitalier de Morlaix, Morlaix

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement

REFERENCES:
- [Background] Hipolito N, Martins S, Ruivo A, Flora S, Silva CG, Marques A, Brooks D, Cruz J. Construct validity and reliability of the Informal Caregiver Burden Assessment Questionnaire (QASCI) in caregivers of patients with COPD. Respir Med. 2022 Dec;205:107027. doi: 10.1016/j.rmed.2022.107027. Epub 2022 Oct 31. PMID 36343503